CLINICAL TRIAL: NCT04495985
Title: Breast Uptake on Radioiodine Scan and Serum Prolactin in Thyroid Cancer Patients Prepared by Thyroid Hormone Withdrawal or Recombinant Human Thyrotropin: A Prospective Study
Brief Title: CASE 1320: RAI Uptake and Serum Prolactin in Thyroid Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 20-488
Record Dates: First submitted 2020-06-10; First posted 2020-08-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thyrogen (rh-TSH): Group 1: Female patients prepared for radioactive iodine treatment by rh-TSH (Thyrogen)
- Withdrawal from thyroid hormone: Group 2: Female patients prepared for radioactive iodine treatment by withdrawal from thyroid hormones

SUMMARY:
Radioactive iodine (RAI) is a radioisotope used to ablate thyroid gland remnant after thyroidectomy in patients diagnosed with differentiated thyroid carcinoma (DTC). A whole body scan (WBS) is performed to not only evaluate for iodine uptake by the native thyroid tissue but also to observe for uptake in other areas of the body, which could be physiological or indicative of iodide-avid metastases. Research has shown a correlation between breast cancer and thyroid cancer. Patients with DTC have been found to have elevated levels of serum prolactin, which could lead to mammary gland dysfunction.

In patients with DTC undergoing RAI scanning or therapy, it has been previously observed that patients prepared by thyroid hormone withdrawal have significantly higher breast uptake on whole body scan compared to those prepared by rh-TSH. Considering the impact of prolactin on breast tissue, this study aims to correlate these findings with the lab values and the method of preparation.

Accordingly, the research question is as follows: does the method of WBS preparation impact prolactin levels and how does that correlate with breast uptake in patients with DTC undergoing RAI WBS?

DETAILED DESCRIPTION:
Radioactive iodine (RAI) is a radioisotope used to ablate thyroid gland remnant after thyroidectomy in patients diagnosed with differentiated thyroid carcinoma (DTC). A whole body scan (WBS) is performed to not only evaluate for iodine uptake by the native thyroid tissue but also to observe for uptake in other areas of the body, which could be physiological or indicative of iodide-avid metastases. Research has shown a correlation between breast cancer and thyroid cancer. Patients with DTC have been found to have elevated levels of serum prolactin, which could lead to mammary gland dysfunction. As such, this study will evaluate for breast uptake on the RAI WBS. Research has shown that patients with DTC may have uptake on RAI WBS.

There is a concern in the molecular imaging community and oncology community that increased I-131 retention in breast tissue may increase the risk of future breast malignancy. The notion that increased serum prolactin concentration increases iodine uptake in breast tissue comes mostly from case series. A correlation between high prolactin as a result of withdrawal from thyroid hormone treatment vs stimulation by recombinant human thyrotropin and uptake by thyroid tissue is the main research question. This research will not be able to answer the question of whether such breast uptake is associated with the future risk breast malignancy. The later research question should be undertaken by other researchers in a larger study with longer follow up. Metastases to the breast from thyroid cancer are rare. Uptake in a discrete lesion in the breast will need to be investigated. It is unclear whether breast adenocarcinoma will concentrate iodine.

In a previous retrospective study of 194 patients with DTC and no breast cancer, it was demonstrated that patients prepared by withdrawal from thyroid hormone had 5-fold higher peak I-131 uptake in breast tissue on post-therapy scan compared to patients prepared by recombinant human thyrotropin (rh-TSH). In other research, DTC patients with hyperprolactinemia have been found to have increased uptake by the mammary gland. The hypothesis is that patients prepared by withdrawal would have increased serum prolactin compared to patients prepared by rh-TSH who are not made hypothyroid. This study plans to prospectively evaluate serum prolactin and breast uptake on the RAI WBS and assess the impact of pre-scan preparation on those variables. This would be the first prospective study of its kind in this set of patients to look at whether the method of pre-RAI scan preparation might impact RAI uptake with correlation to prolactin levels.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with diagnosis of differentiated thyroid carcinoma who have had thyroidectomy performed previously
* Patients able to understand and sign informed consent for imaging
* Patients already scheduled to undergo radioactive iodine whole body scanning (RAI WBS)

Exclusion Criteria:

* Males
* Patients with a history of breast cancer
* Patients with a known history of hyperprolactinemia
* Patients receiving medications known to raise serum prolactin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Female patients with differential thyroid cancer prepared for radioactive iodine whole body scan by withdrawal from thyroid hormones Group 2: Female patients with differential thyroid cancer prepared for radioactive iodine whole body scan by rh-TSH.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Breast uptake of I-131 on whole body radioactive iodine scan | 10 days after treatment
  Breast uptake of I-131 on whole body radioactive iodine scan

SECONDARY OUTCOMES:
Change in serum prolactin concentration | 6 weeks
  Change in prolactin levels in thyroid hormone withdrawal group
Serum prolactin concentration | 3 days
  Change in prolactin levels in thyrogen preparation group
Prolactin level and breast uptake of I-131 | Day 46 of thyroid hormone withdrawal group
  Correlation between serum prolactin level and breast uptake of I-131
Prolactin level and breast uptake of I-131 | Day 26 of thyrogen preparation group
  Correlation between serum prolactin level and breast uptake of I-131

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Mikhael, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No